CLINICAL TRIAL: NCT00188526
Title: CT Guided Lung Biopsy: Core or Fine Needle Aspiration
Brief Title: Computed Tomography (CT) Guided Lung Biopsy: Core or Fine Needle Aspiration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unknown Reason
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-0516
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: lung biopsy

SUMMARY:
This study is a comparison of core needle biopsy with fine needle aspiration biopsy in the evaluation of lung nodules.

ELIGIBILITY:
Inclusion Criteria:

* All patients having a lung biopsy

Exclusion Criteria:

* Lymphoma

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Study Completion 2006-09

PRIMARY OUTCOMES:
Diagnostic accuracy

SECONDARY OUTCOMES:
Complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, FRCP C, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada